CLINICAL TRIAL: NCT02110212
Title: A Prospective, Randomized Study of Cataract Surgery With the Assistance of the OptiMedica Femtosecond Laser System Compared to Standard Surgical Procedure of Continuous Curvilinear Capsulorhexis and Ultrasonic Phacoemulsification
Brief Title: Femtosecond Laser for Cataract Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA approval received for product, no additional study subjects required.
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMC-C-3.0
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: Cataract; Surgery, cataract extraction; Optical devices, laser
MeSH Terms: conditions — Cataract | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- U/S Surgery and CCC (Active Comparator): Ultrasound (U/S) cataract surgery and continuous curvilinear capsulorhexis (CCC).
  Interventions: Procedure: U/S Surgery and CCC
- FS Laser Surgery (Experimental): For femtosecond laser-assisted cataract surgery (FS Laser Surgery), subjects will receive capsulotomy, lens segmentation and, at investigator discretion, lens softening using the femtosecond laser device.
  Interventions: Device: FS Laser Surgery

INTERVENTIONS:
Procedure: U/S Surgery and CCC — Subjects will receive the standard of care for U/S cataract surgery and CCC to facilitate removal of the crystalline lens.
  Other Names: Standard of care for U/S and CCC was required.
  Arms: U/S Surgery and CCC
Device: FS Laser Surgery — The Catalys System is an ophthalmic surgical laser system intended for use in cataract surgery.
  Other Names: OptiMedica Catalys™ Precision Laser System (Catalys System)
  Arms: FS Laser Surgery

SUMMARY:
The objective of this study is to evaluate the safety and efficacy the OptiMedica Femtosecond Laser System, also known as the Catalys™ Precision Laser System, to perform two surgical maneuvers used in the treatment of subjects with cataracts. Efficacy will be evaluated by comparisons to the standard surgical procedure of continuous curvilinear capsulorhexis (CCC) and ultrasonic phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the treatment/follow-up schedule and requirements
* Able to understand and provide written Informed Consent
* ETDRS visual acuity equal to or worse than 20/32 (best corrected)
* Age between 50 and 80 years old
* Pupil dilates to at least 6 mm
* Subject able to fixate
* Grade 1-4 nuclear sclerotic cataract (LOCS III)
* Axial length between 22 and 26 mm

Exclusion Criteria:

* Pregnant, intending to become pregnant during course of the study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
* Participation in a study of another device or drug within 3 months prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria
* Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study or for which cataract surgery is contraindicated
* Anterior chamber depth (anterior corneal surface to anterior capsule margin) less than 2.5 mm via IOL Master (Zeiss).
* History of prior ocular surgery
* History of ocular trauma
* Co-existing ocular disease affecting vision
* History or current use of alpha-1 antagonist medication (e.g., Flomax)
* Known sensitivity to planned concomitant medications

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Capsulotomy Dimension | Day of Surgery
  Capsulotomy size will be measured during surgery for both the experimental and control groups.

SECONDARY OUTCOMES:
Cumulative Dissipated Energy (CDE) | Day of Surgery
  CDE (the amount of ultrasound energy delivered during phacoemulsification of the crystalline lens) used will be measured during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Batlle, MD, Principal Investigator — Laser Center; William W. Culbertson, MD, Study Director — Bascom Palmer Eye Institute